CLINICAL TRIAL: NCT03235375
Title: A Phase 1, Open-Label, Single Dose, Parallel-Group Study to Evaluate the Pharmacokinetics, Safety and Tolerability of MEDI0382 in Subjects With Renal Impairment
Brief Title: A Study to Evaluate Pharmacokinetics, Safety and Tolerability of MEDI0382 in Renal Impairment Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D5670C00008
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Renal Insufficiency
Keywords: Kidney Failure, Kidney Insufficiency, Renal Failure, Renal Insufficiency, MEDI0382
MeSH Terms: conditions — Renal Insufficiency | interventions — cotadutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: End Stage Renal Disease (ESRD) (Experimental): Subjects with CrCl <20ml/min will receive MEDI0382 administered subcutaneously
  Interventions: Drug: MEDI0382
- Group 2: Severe and ESRD Subjects (Experimental): Subjects with CrCl >20 and < 30 ml/min will receive MEDI0382 administered subcutaneously
  Interventions: Drug: MEDI0382
- Group 3: Healthy Subjects (Active Comparator): Subjects with CrCl >90 ml/min will receive MEDI0382 administered subcutaneously
  Interventions: Drug: MEDI0382
- Group 4: Moderate Renal Disease (Experimental): Subjects with CrCl > or equal to 30 and < 60 mL/min will receive MEDI0382 administered subcutaneously
  Interventions: Drug: MEDI0382

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 administered subcutaneously

SUMMARY:
A phase 1 open-label, single-dose study to evaluate the pharmacokinetics (PK), safety, tolerability and immunogenicity of MEDI0382 in subjects with renal impairment.

DETAILED DESCRIPTION:
This is an open-label, single-dose, parallel group study to evaluate the PK, safety, tolerability, and immunogenicity of MEDI0382 in subjects with renal impairment. Enrollment of approximately 40 subjects across multiple sites is planned. Subjects will be divided into 4 groups based on renal function.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent
* BMI greater than or equal to 17 and less than or equal to 40 kg/m2
* Creatinine clearance rate greater than or equal to 90 (healthy); or renally impaired (less than 60 mL/min)
* Females of childbearing potential must use a highly effective form of contraception.

Exclusion Criteria:

* Any history of or concurrent condition that in the opinion of the investigator would compromise the subjects safety.
* Subjects on dialysis
* Subjects with pancreatitis
* Renal transplant subjects
* Females pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration of MEDI0382 (Cmax) | 0-48 hours
  The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data
Area under the Concentration Time Curve (AUC) of MEDI0382 | 0-48 hours
  The area under the plasma concentration-time curve to 48 hours concentration determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations

SECONDARY OUTCOMES:
Time to maximum observed concentration (Tmax) | 0-48 hours
  Time to maximum observed concentration.
apparent clearance (Cl/F) | 0-48 hours
  The apparent clearance will be calculated as CL/F=Dose/AUC(0-inf)
AUCinf | 0-48 hours
  The AUC extrapolated to infinity will be calculated, where data permit, as the sum of AUC((0-t) and Ct/z, where Ct is the observed plasma concentration obtained from the log-linear regression analysis of the last quantifiable time-point and z is the terminal phase rate constant.
Half-life (T1/2) | 0-48 hours
  The apparent terminal elimination half-life (t1/2) obtained as the ratio of ln2/z, where z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data
Anti-drug Antibody (ADA) titer | Day -1 to day 28
  ADA titer through to day 28
Number of subjects with Adverse Events | Study onset till 28 days post dosing
  Treatment emergent adverse events (TEAEs) and serious adverse events (TESAEs)
Number of subjects with Adverse Events | Study onset till 28 days post dosing
  Vital Signs (systolic and diastolic blood pressure, pulse rate, temperature and respiratory rates)
Number of subjects with Adverse Events | Study onset till 28 days post dosing
  Clinical laboratory assessments (serum chemistry, hematology, and urinalysis)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (2):
  - Research Site, Kiel
  - Research Site, München
- New Zealand (2):
  - Research Site, Auckland
  - Research Site, Christchurch

REFERENCES:
- [Derived] Klein G, Petrone M, Yang Y, Hoang T, Hazlett S, Hansen L, Flor A. Pharmacokinetics and Safety of Cotadutide, a GLP-1 and Glucagon Receptor Dual Agonist, in Individuals with Renal Impairment: A Single-Dose, Phase I, Bridging Study. Clin Pharmacokinet. 2023 Jun;62(6):881-890. doi: 10.1007/s40262-023-01239-1. Epub 2023 May 4. PMID 37140727